CLINICAL TRIAL: NCT00937027
Title: A Randomized Phase 1 Study Comparing The Safety and Oral Pharmacokinetics Of 0.25 mg and 1.0 mg Aminopterin Tablets In Human Subjects With Psoriasis
Brief Title: Aminopterin Pharmacokinetic Study In Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Syntrix-AMT-PSO-101; NIH Grant #: R43AI068282
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2012-11

CONDITIONS: Psoriasis
Keywords: Antifolate; Psoriasis; Antiinflammatory drug; Autoimmune disease; Treatment
MeSH Terms: conditions — Psoriasis; Autoimmune Diseases | interventions — Aminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminopterin one 1.0 mg tablet (Active Comparator)
  Interventions: Drug: Aminopterin
- Aminopterin 1 four 0.25 mg tablets (Active Comparator)
  Interventions: Drug: Aminopterin

INTERVENTIONS:
Drug: Aminopterin — oral tablets, 1.0 mg dose, once weekly, two weeks

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic properties (the absorption, distribution and excretion) of two preparations of aminopterin (0.25 mg tablets and 1.0 mg tablets) following oral administration by subjects with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent by signing an IRB-approved Informed Consent.
* Be under treatment for at least moderate to severe psoriasis (diagnosis confirmed by a dermatologist) with MTX (10-20 mg per week) for a minimum of 3 months. Moderate to severe psoriasis is defined here as plaque-type psoriasis affecting a body surface area > 10%.
* Be 21 years of age or older, but not 60 years of age or older.
* If participant is female of child bearing potential, then subject must indicate that she is not pregnant.
* Must be fully informed of the potential for AMT to adversely affect a fetus, and must agree to use highly effective method of birth control beginning at the time of consent, during the study, and for 3 months after leaving the study.
* Women of childbearing potential may enter the study only after a confirmed menstrual period, and must have a negative urine pregnancy test at the time of screening and within 24 hours of each study drug dose.
* Have adequate hematologic function as evidenced by the following :results obtained from a blood sample drawn within 2 days of day 0:

  * WBC > 4,500/ mm3
  * Platelet Count > 150,000/mm3
  * Hemoglobin > 12.0 gm/dL
* Have adequate liver function as evidenced by the following results obtained from a blood sample drawn within 2 days of day 0:

  * AST (SGOT) ≤ 40 IU/L
  * ALT (SGPT) ≤ 40 IU/L
  * Alkaline Phosphatase ≤ 120 IU/L
  * Total Bilirubin ≤ 1.2 mg/dL
* Have adequate renal function as evidenced by the following result obtained from a blood sample drawn within 2 days of day 0:

  * GFR estimated by Cockcroft-Gault formula:
  * > 90 ml/min (male)
  * > 90 ml/min (female)
* Have no detectable urine glucose, urine ketones, or urine protein from a sample obtained within 2 days of day 0.
* Weight of 35 to 90 kg.

Exclusion Criteria:

* A known history of hepatitis, liver fibrosis or cirrhosis (grades IIIA, IIIB or IV), diabetes (type I or II), HIV infection, tuberculosis, interstitial lung disease, or an abnormal screening chest x-ray that is consistent with interstitial lung disease.
* Known peptic ulcer, ulcerative colitis or Crohn's disease.
* Body mass index (BMI) <19.0 or > 35.0 (see appendix C).
* Within 2 weeks prior to randomization use of any of the following medications that may result in drug/drug interactions with aminopterin: methotrexate, trimethoprim with or without sulfamethoxazole; sulfonamides; sulfonylureas; pyrimethamine; triamethamine; dipyridamole; colchicine; probenecid; aminoglycosides; theophylline; phenytoin; and folinic acid (i.e., leucovorin) unless prescribed by the investigator to treat study drug related toxicity.
* Within 2 weeks prior to randomization use of salicylates, non-steroidal anti-inflammatory (NSAID) drugs, including Over-The-Counter nonprescription use of aspirin, ibuprofen or naproxen.
* Use of medications that may be negatively influenced by regular folic acid supplementation such as the anti-epileptics phenobarbital, diphenylhydantoin, and primidone.
* Use of any investigational medication within 30 days prior to admission to the study.
* Inability to abstain from alcohol during the study.
* A history of substance abuse, drug addiction or alcoholism.
* Unwillingness to use an adequate form of contraception during the study and for 3 months after the study.
* A female who is pregnant, intends to become pregnant during the study (or within 6 months after study completion), or nursing.
* Concurrent participation in another clinical trial involving experimental treatment.
* Current and uncontrolled infection, cardiovascular, pulmonary, hepatic or GI conditions that will interfere with the conduct of the trial or pose an additional morbid risk.
* Any renal conditions that will interfere with the conduct of the trial or pose an additional morbid risk.
* Any concurrent disease or condition that in the opinion of the investigator impairs the subject's ability to complete the trial. Psychological, familial, sociological, geographical or medical conditions which, in the Investigator's opinion, could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial's data.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Aminopterin area under the curve | 0.0, 0.5, 1.0, 1.5, 2.0, 3.0, 5.0, 7.0, 10.0 and 12.0 hours
Adverse events | 14 days

SECONDARY OUTCOMES:
Aminopterin concentration maximum, time to maximal aminopterin concentration, aminopterin volume of distribution and aminopterin half-life. | 0.0, 0.5, 1.0, 1.5, 2.0, 3.0, 5.0, 7.0, 10.0 and 12.0 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alan Menter, M.D., Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States

REFERENCES:
- [Derived] Menter A, Thrash B, Cherian C, Matherly LH, Wang L, Gangjee A, Morgan JR, Maeda DY, Schuler AD, Kahn SJ, Zebala JA. Intestinal transport of aminopterin enantiomers in dogs and humans with psoriasis is stereoselective: evidence for a mechanism involving the proton-coupled folate transporter. J Pharmacol Exp Ther. 2012 Sep;342(3):696-708. doi: 10.1124/jpet.112.195479. Epub 2012 May 31. PMID 22653877